CLINICAL TRIAL: NCT04410081
Title: An Open-Label Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-JNJ-73841937 (Lazertinib) After a Single Oral Dose in Healthy Male Participants
Brief Title: A Study of (14C)-JNJ-73841937 (Lazertinib) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR108791; 73841937NSC1004 (Other: Janssen Research & Development, LLC); 2020-000646-34 (EudraCT Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 14C-lazertinib (Experimental): Participants will receive a single oral dose of 14C-lazertinib on Day 1.
  Interventions: Drug: 14C-lazertinib

INTERVENTIONS:
Drug: 14C-lazertinib — A single oral dose of 14C-lazertinib will be administered.
  Other Names: JNJ-73841937

SUMMARY:
The purpose of this study is to characterize the absorption, metabolic pathways of lazertinib, and the excretion of the parent lazertinib and its metabolites, after a single oral dose of 14C-lazertinib in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of medical history performed at screening and physical examination and vital signs (pulse rate and body temperature) performed at screening and admission to the study site
* Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry or hematology panel are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2, inclusive (BMI = weight/height^2), and body weight not less than 50 kg at screening
* Blood pressure at screening and admission to the study site (after the participant supine for 5 minutes) between 90 and 140 millimeter of Mercury (mmHg) systolic, inclusive; and no higher than 90 mmHg diastolic at screening
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, including: Sinus rhythm, Pulse rate between 45 and 100 beats per minute (bpm), corrected QT (QTc) interval less than or equal to (<=) 450 millisecond (msec), QRS interval of less than (<)120 msec, PR interval <210 msec

Exclusion Criteria:

* History of infection suspected or confirmed to be related to Coronavirus disease 2019 (COVID-19) within 4 weeks before intake of study drug
* Participant has known allergies, hypersensitivity, or intolerance to lazertinib or any of its excipients
* Participant has a positive test for hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen (HBsAg), hepatitis B (anti-HBc or anti-HBs), or hepatitis C (anti-HCV) antibodies positive at screening. Hepatitis B surface antibody positivity is not exclusionary if participant can provide evidence of Hepatitis B vaccination
* Participant who plans to father a child while enrolled in the study or within 6 months after study drug administration
* Exposure to radiation for professional or medical reasons with the exception of up to 2 standard diagnostic radiographs (example, [dental X-rays, plain chest X-ray]) within 1 year before study drug administration on Study Day 1. Participants cannot have participated in a radiolabeled drug study within 12 months prior to dosing if the dose was higher than 0.1 megabecquerel (MBq)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of 14C-lazertinib | Up to 99 days
  Cmax is defined as maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of 14C-lazertinib | Up to 99 days
  Tmax is defined time to reach the maximum observed concentration.
Area Under the Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUC [0-last]) of 14C-lazertinib | Up to 99 days
  AUC (0-last) is defined as area under the plasma concentration-time curve from time 0 to the time of last observed quantifiable concentration.
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of 14C-lazertinib | Up to 99 days
  AUC (0-infinity) is defined as area under the plasma concentration-time curve from time 0 to infinity, calculated as the sum of AUC(0-last)+C(last)/ lambda(z), where C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Half-life (t1/2) of 14C-lazertinib | Up to 99 days
  Elimination half-life associated with the terminal slope lambda(z) of the semilogarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Apparent Terminal Elimination Rate Constant (Lambda[z]) | Up to 99 days
  Lambda(z) is defined as apparent terminal elimination rate constant, estimated by linear regression using the terminal log-linear phase of the log transformed concentration vs time data.
Total Apparent Clearance (CL/F) of 14C-lazertinib | Up to 99 days
  Clearance is a quantitative measure of the rate at which a drug substance is removed from the body, calculated as dose/AUC (0-infinity).
Apparent Volume of Distribution (Vdz/F) of 14C-lazertinib | Up to 99 days
  Apparent volume of distribution, calculated as dose/(Lambda(z)*AUC (0-infinity).
Ratio of Blood to Plasma Total Radioactivity of 14C-lazertinib | Up to 99 days
  Blood to plasma total radioactivity ratio, calculated as blood total radioactivity/plasma total radioactivity.
Ratio of AUC (0-infinity) of 14C-lazertinib to AUC (0-infinity) of Total Radioactivity in Plasma | Up to 99 days
  The ratio of AUC (0-infinity) of 14C-lazertinib to AUC (0-infinity) of total radioactivity in plasma will be assessed.
Ratio of AUC (0-last) of 14C-lazertinib Concentration to AUC (0-last) of Total Radioactivity in Plasma | Up to 99 days
  The ratio of AUC (0-last) of 14C-lazertinib to AUC (0-last) of total radioactivity in plasma will be assessed.
Ratio of Cmax of 14C-lazertinib to Cmax of Total Radioactivity in Plasma | Up to 99 days
  The ratio of Cmax of 14C-lazertinib to Cmax of total radioactivity in plasma will be assessed.
Ratio of 14C-lazertinib Concentration to Total Radioactivity in Plasma | Up to 99 days
  The ratio of 14C-lazertinib concentration to total radioactivity in plasma for each sampling time point will be assessed.
Amount of 14C-lazertinib Excreted in Urine (Ae[t1-t2]) | Up to 99 days
  Amount excreted into the urine during a collection interval, where t1 and t2 are the start and end times of the collection interval, and calculated by multiplying the urinary volume with the urinary concentration for that interval.
Cumulative Amount of 14C-lazertinib Excreted in Urine (Ae) | Up to 99 days
  Cumulative amount excreted into the urine over the entire collection period, calculated as the sum of Ae's across the collection intervals for each participant.
Percentage of 14C-lazertinib Dose Excreted in Urine (%Ae) | Up to 99 days
  Cumulative amount excreted into the urine, expressed as a percentage of the administered dose, calculated as (Ae divided by dose)*100.
Renal Clearance (CLr) of 14C-lazertinib | Up to 99 days
  The CLr is the renal clearance of the drug, calculated as Ae/AUC(0-infinity).
Amount of 14C-lazertinib Excreted in Feces (Fe[t1-t2]) | Up to 99 days
  Amount excreted into the feces during a collection interval, where t1 and t2 are the start and end times of the collection interval, and calculated by multiplying the feces weight with the feces concentration for that interval.
Cumulative Amount of 14C-lazertinib Excreted in Feces (Fe) | Up to 99 days
  Cumulative amount excreted into the feces over the entire collection period, calculated as the sum of Fe's across the collection intervals for each participant.
Percentage of 14C-lazertinib Dose Excreted in Feces (%Fe) | Up to 99 days
  Cumulative amount excreted into the feces, expressed as a percentage of the administered dose, calculated as (Fe divided by dose)*100.
Total Recovery of 14C-lazertinib Dose in Feces and Urine | Up to 99 days
  Total recovery, calculated as sum of %Ae and %Fe.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 135 days
  An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency